CLINICAL TRIAL: NCT00066014
Title: Clinical Investigation of Mandibular Implant Overdenture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIDCR-12204; R01DE012204 (NIH); NCT00000366 (obsolete NCT alias)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2010-01

CONDITIONS: Dental Implantation
Keywords: Dental Implantation-Osseointegrated; Dentures; Dental Prostheses; Denture, Implant-Supported

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment modalities changed for comparison (Active Comparator): All subjects experienced all treatment modalities being studied.
  Interventions: Procedure: Implant Overdenture Treatment

INTERVENTIONS:
Procedure: Implant Overdenture Treatment — All overdenture treatment modalities were provided to each subject using a crossover design.

SUMMARY:
The purpose of this study is to compare the effectiveness of three variable dental implant attachment methodologies in conjunction with lower dental-implant retained/supported complete overdenture treatment. These three methods are all presently used by dental practitioners, but vary significantly in terms of added treatment cost and complexity. The study tests the hypothesis that the least complex and costly method provides an equivalent treatment outcome to other more complex and costly methods.

DETAILED DESCRIPTION:
This project utilizes 30 subjects in a prospective, randomly assigned clinical study that uses a four-period, six sequence, three treatment crossover design to test the hypothesis that defined outcomes of variable implant overdenture treatments are equivalent. The project tests three overdenture treatment modalities, (1) four-implant, bar/clip-attached treatment, (2) two-implant, bar/clip-attached treatment, and (3) two-implant independently attached (O-ring) treatment. Each subject has four dental implants placed into the anterior mandible and new dentures are fabricated. After successful implant integration, subjects are randomly assigned to one of six sequences of treatment. Each treatment is followed for data collection for at least twelve months before the mandibular denture is modified to incorporate the next treatment in the sequence. Equivalence is measured in terms of prosthesis retention, stability, supporting and peri-implant tissue response, patient satisfaction/preference and treatment complications/failures.

Information from this study will assist dental practitioners during treatment planning in selecting appropriate and cost effective treatment choices. There is an inverse relationship between edentulism in the U.S. population and socioeconomic status. If less costly and simplified treatment methods are shown to provide an equivalent treatment outcome to more costly/complex methods, these simplified treatments can be used to treat a larger percentage of the edentulous population.

ELIGIBILITY:
Inclusion:

* Adult patient;
* Male or female;
* At least one year of previous conventional complete denture treatment history;
* Willing to accept the conditions of the study and informed consent freely given;
* Ability to participate for 6 years;
* Able to understand and respond to self-reporting measurement scales used in the study;
* Minimum 20-mm interarch distance at the estimated vertical dimension of occlusion;
* Adequate bone quality;
* Adequate bone quantity to accommodate minimally four 3.75-mm diameter by 7-mm long Brånemark implants.

Exclusion:

* Administrative or physical considerations which would seriously affect the surgical procedure or construe a hindrance for a six-year involvement;
* History of drug or alcohol abuse;
* Excessive smoking (1+ pack/day);
* Uncontrolled systemic disease;
* Inability to undergo minor oral surgery because of health or personal reasons;
* Irradiated surgical site;
* Unrealistic expectations of the prosthodontic treatment outcome;
* Psychological or psychiatric conditions that could influence the subject's reaction to treatment;
* Acute or chronic TMD problems;
* pregnancy;
* Class II jaw relationship;
* Conventional dental treatment the treatment of choice.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Comparison of implant overdenture clinical modalities using clinical measures to compare treatment outcomes | 6 month and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: David R Burns, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States